CLINICAL TRIAL: NCT02977078
Title: Improving Asthma Treatment Using Inhaler Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 14RM008; 193750 (Other: IRAS)
Record Dates: First submitted 2016-11-18; First posted 2016-11-30 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Asthma
Keywords: Inhaler
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Sham Comparator): Inhaler use monitored by device but no feedback to participants (control); this group is unaware of the second arm receiving feedback on inhaler use.
  Interventions: Device: Inhaler casing
- Active (Experimental): Inhaler use monitored with feedback to participants (active); participants randomized to this group sign an additional consent to receive feedback on inhaler use
  Interventions: Behavioral: Active feedback on monitored inhaler use; Device: Inhaler casing; Device: Mobile application

INTERVENTIONS:
Behavioral: Active feedback on monitored inhaler use — Feedback given on inhaler use by research nurse/ doctor based on mobile application feedback
  Arms: Active
Device: Inhaler casing — Monitors inhaler use
Device: Mobile application — Mobile application software linked to inhaler casing
  Arms: Active

SUMMARY:
This study will use inhaler technology to observe and feedback overall patterns of medication use. We will look at whether this improves preventer inhaler use and reduces reliever inhaler overuse.

We will also assess whether inhaler technology is patient-friendly and cost effective, whether it helps with treatment decisions in asthma and whether it can help us to predict and prevent asthma attacks.

DETAILED DESCRIPTION:
The SmartTouch™ range of electronic casings will record the use of metered dose inhalers (MDI) by participants in the study. The actuation data can be remotely viewed and analyzed by the investigators.

The hypothesis is that employing such technology to measure medication patterns and to help provide patient feedback improves inhaler adherence and potentially clinical outcomes (asthma control and exacerbations) in asthma patients with recent asthma attacks in a practical, real-world setting.

We will assess whether electronic inhaler data capture can identify patients requiring more frequent reviews or treatment change and enable proactive self- management.

Using qualitative methods, we will explore participants' attitudes to their asthma management, whether the use of inhaler technology has had an impact on this and whether they found its use acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Use of systemic corticosteroids for worsening asthma (or an increase from baseline dose in patients on long-term oral corticosteroids) in the prior 12 months [i.e. at least one asthma exacerbation requiring additional systemic corticosteroid in the prior 12 months] patient reported.
* Doctor's diagnosis of asthma for at least 12 months
* On BTS step 2-5 treatment via MDI [monitoring devices to be utilised in the study are compatible with MDI inhalers]
* Use of own internet-enabled and compatible mobile phone

Exclusion Criteria:

* Diagnosis of COPD or onset of symptoms after the age of 40 in patients with ≥10 Pack Year History of smoking
* Other clinically significant coexisting respiratory disease e.g. fibrosis, bronchiectasis
* Patients on maintenance and reliever therapy ('SMART' or 'Fostair® MART')

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Impact on adherence to preventative medication use based on the mean percentage of prescribed doses taken daily over the study period | Upto 24 weeks (study duration)
  Co-primary endpoint
Impact on adherence to reliever medication use based on the number of days with >16 actuations/day of Salbutamol taken in a 24-hour period | Upto 24 weeks (study duration)
  Co-primary endpoint

SECONDARY OUTCOMES:
Patient acceptability via qualitative feedback with questionnaires | Upto 24 weeks (study duration)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Shaw, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Queens Medical Centre Campus, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Adejumo I, Patel M, McKeever TM, Shaw DE. Does inhaler technology improve adherence and asthma control? A pilot randomized controlled trial. Ann Allergy Asthma Immunol. 2022 Jun;128(6):727-729. doi: 10.1016/j.anai.2022.02.023. Epub 2022 Mar 4. No abstract available. PMID 35257874